CLINICAL TRIAL: NCT04613466
Title: The Prevelance of Pulmonary Manifestations in Patients With Inflammatory Bowel Disease
Brief Title: The Prevelance of Pulmonary Manifestation in Patients With Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hayam Fathy Nasr, clinical doctor of internal medicine, Assiut University
Other Study IDs: Gateroentrolgy unit
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: The Prevelance and Complications of Pulmonary Manifestations in Patients With Inflammatory Bowel Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bronchopulmonary manifestations signs and symptoms are variable extraintestinal manifestations of IBD.

DETAILED DESCRIPTION:
Several cases like bronchiactsis, bronchitis, tracheobronchitis and broncholitis. None of this complications are specific for either crohns or ulcerative , however the majority of cases are related to ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:All patients diagnosed ulcerative colitis and crohns disaese on conventional treatment and biological treatment -

Exclusion Criteria:no exclusion criteria

-

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Gender Based: Yes — rural or urban
Study Population: All patients diagnosed IBD either male or female age 18 to 60 years
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The presence of pulmonary manifestations in IBD patients | 1 year